CLINICAL TRIAL: NCT03671720
Title: Personalized Vaccine Generated by Autologous Dendritic Cells Pulsed With Autologous Whole Tumor Cell Lysate Treat Advanced Solid Tumor Patients With High Tumor Mutation Burden
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Capital Medical University (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Jun Ren MD, PhD, Director of Captial Medical University Cancer Center, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCL DC Vaccine for TMB-High
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- personalized vaccine (Experimental)
  Interventions: Biological: personalized DC vaccine

INTERVENTIONS:
Biological: personalized DC vaccine — personalized vaccine comprised of autologous dendritic cells (DC) loaded in vitro with lysate from autologous tumor cells, administered intranodally on day 1,8,15, with a combination of oral cyclophosphamide (50mg) every day except the day of vaccine administrations.Cycles are repeated every 21 days. Treatment is continued until disease progression or exhaustion of vaccine supply, whichever comes first.

SUMMARY:
The study is to investigate the safety and efficacy of dendritic cells vaccines pulsed with autologous whole tumor cell lysate for treating advanced solid tumor patients with high tumor mutation burden.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced or metastatic solid tumors.
2. Patients must have received previously standard therapy for that malignancy or declined to chemotherapy/radiotherapy.
3. Estimated life expectancy > 3 months
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2.
5. Age 18~75 years old
6. Next-generation sequencing identified tumor mutation burden higher than 9 Muts/MB in tumor tissue or peripheral blood samples.
7. Available for the adequate surgical or core-needle biopsy specimens from primary or metastasis lesions to manufacture the DC vaccines.
8. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
9. Adequate hematologic function, with WBC ≥ 3000/microliter, hemoglobin ≥ 9 g/dL (it is acceptable to have had prior transfusion), platelets ≥ 75,000/microliter; PT-INR <1.5 (unless patient is receiving warfarin in which case PT-INR must be <3), PTT <1.5X ULN
10. Adequate renal and hepatic function, with serum creatinine < 1.5 mg/dL, bilirubin < 1.5 mg/dL (except for Gilbert's syndrome which will allow bilirubin ≤ 2.0 mg/dL), ALT and AST ≤ 2.5 x upper limit of normal.

Exclusion Criteria:

1. Patients with a history of autoimmune disease, such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. Autoimmune related thyroid disease and vitiligo are permitted.
2. Patients with serious intercurrent chronic or acute illness, such as cardiac disease (NYHA class III or IV), hepatic disease, or other illness considered by the Principal Investigator as unwarranted high risk for investigational drug treatment.
3. Patients with a medical or psychological impediment to probable compliance with the protocol should be excluded.
4. Concurrent (or within the last 5 years) second malignancy other than non melanoma skin cancer, cervical carcinoma in situ, controlled superficial bladder cancer, or other carcinoma in situ that has been treated.
5. Presence of an active acute or chronic infection including: a urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot). Patients with HIV are excluded based on immuno-suppression, which may render them unable to respond to the vaccine; patients with chronic hepatitis are excluded because of concern that hepatitis could be exacerbated by the injections.
6. Patients on chronic steroid therapy (or other immuno-suppressives, such as azathioprine or cyclosporin A) are excluded on the basis of potential immune suppression. Patients must have had 6 weeks of discontinuation of any steroid therapy (except that used as pre-medication for chemotherapy or contrast-enhanced studies or for acute treatment (<5 days) of intercurrent medical condition such as a gout flare) prior to enrollment.
7. Pregnant and nursing women should be excluded from the protocol since this research may have unknown and harmful effects on an unborn child or on young children. If the patient is sexually active, the patient must agree to use a medically acceptable form of birth control while receiving treatment and for a period of 4 months following the last vaccination therapy. It is not known whether the treatment used in this study could affect the sperm and could potentially harm a child that may be fathered while on this study.
8. Patients with acute or chronic skin disorders that will interfere with injection into the skin of the extremities or subsequent assessment of potential skin reactions will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Treatment-related adverse events | 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.All toxicities observed within 30 days of last vaccination will be included.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 6 months
  The rate of patients was evaluated as complete response or partial response
Progression-free survival of the participants(PFS) | 24 months
  From starting date of vaccine treatment until date of first documented disease progression or date of death from any cause, whichever comes first
Overall survival of the participants(OS) | 24 months
  From starting date of vaccine treatment until date of death from any cause
The changes in immune-response specific patient-reported outcomes(irPRO) | 24 months
  To assess the irPRO scale ratings prior to and after the cancer immunotherapy
The changes in patient self-reported quality of life | 24 months
  To assess the EORTC QLQ-C30 scale ratings prior to and after the cancer immunotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University Cancer Center/Beijing Shijitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No